CLINICAL TRIAL: NCT02792504
Title: POST MARKETING SURVEILLANCE TO OBSERVE THE SAFETY AND EFFICACY OF DUAVIVE TAB 0.45MG/20MG
Brief Title: Post Marketing Surveillance To Observe Safety And Efficacy Of Duavive
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B2311067
Record Dates: First submitted 2016-02-19; First posted 2016-06-07 (Estimated); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Severe Vasomotor Symptom Associated With Menopause

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate safety and efficacy of CE/BZA in real practice in Korea

ELIGIBILITY:
Inclusion Criteria:

1. Severe post menopausal vasomotor symptoms with uterus
2. postmenopausal osteopenia

Exclusion Criteria:

* Women with undiagnosed abnormal uterine bleeding
* Women with known, suspected, or past history of breast cancer
* Women with known or suspected estrogen-dependent neoplasia
* Women with active deep venous thrombosis, pulmonary embolism, or history of these conditions
* Women with active arterial thromboembolic disease (for example, stroke, myocardial infarction) or history of these conditions
* Women who are receiving progestin, estrogen, or estrogen-agonists/antagonists
* Women with hypersensitivity (for example, anaphylaxis, angioedema) to estrogens, bazedoxifene, or any ingredients
* Women with known hepatic impairment or disease
* Women with known protein C, protein S, or antithrombin deficiency or other known thrombophilic disorders
* Pregnant women, women who may become pregnant, and nursing mothers
* Women with hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose galactose malabsorption.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: General hospital and Primary clinic in Korea
Sampling Method: Probability Sample
Enrollment: 669 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- South Korea (19):
  - Kyungpook National University/Department of Internal Medicine (Cardiology), Jung-gu, Daegu
  - Dr. Wang's OB & GY Clinic, Seoul, Dobong-gu
  - Kimhyeonmi OBGY, Hwaseong-si, Dongtan
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Bucheon St. Mary Hospital The Catholic University of Korea, Bucheon-si, Gyeonggi-do
  - Baylor Ewha Obgyn Clinic, Seongnam-si, Gyeonggi-do
  - Dongguk University Ilsan Medical Center Obstetrics, Goyang-si, Ilsandong-gu
  - Obstetrics / Grace Women's Hospital, Goyong-si, Ilsandong-gu
  - Kyungpook National University Hospital, Obstetrics, Daegu, Jung-gu
  - Pusan University Hospital Obstetrics, Pusan, Seo-gu
  - Catholic Universith of Korea, Seoul ST. Mary's Hospital, Seoul, Seocho-gu
  - Samsung Medical Center, Sungkyunkwan Univ. School of Medicine, Kangnam-ku, Seoul
  - Konkuk University Medical Center, Seoul
  - Seoul National University Hospital / Department of Internal Medicine, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Sanggye Paik Hospital-Inje University, Seoul
  - Chungang University Hospital, Seoul
  - AJOU University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B2311067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study was conducted in Korea. Enrolled participants included were administered with Duavive tablet 0.45 milligram (mg)/20 mg (conjugated estrogens 0.45 mg, bazedoxifene acetate 20 mg) for the first time as a part of routine treatment after the start of the study at a study site and complied with the local labeling. Participants were planned to be evaluated for 3 months, 6 months or more depending upon till when Duavive tablet was administered based on investigator's judgement.
Pre-assignment Details: In this study no screening was performed. Women participants who were administered Duavive tablet were enrolled.
Groups:
- Duavive: Participants were administered with Duavive tablet as part of routine practice in Korean health care centers by accredited physicians per the local product document.
Period: Overall Study
Arm/Group | Duavive
Started | 669
Safety Analysis Set | 639
Efficacy Analysis Set | 390
Completed | 639
Not Completed | 30
Not completed — Lost to Follow-up | 24
Not completed — Violated inclusion/exclusion criteria | 6

BASELINE CHARACTERISTICS:
Population: Safety analysis set included those participants who had been administered with Duavive tablet at least once and had completed follow up.
Arm/Group | Duavive
Number analyzed (Participants) | 639
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.65 (5.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 639
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. AEs included both serious and all non-serious adverse events.
Time Frame: Baseline up to 28 days after last dose of study drug (up to 22 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Duavive
Number analyzed (Participants) | 639
Participants
  AEs | 73
  SAEs | 2

2. Primary Outcome: Number of Participants With Treatment Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. A treatment-related adverse event was any untoward medical occurrence attributed to Duavive tablet in a participant who received Duavive tablet. A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to Duavive tablet was assessed by the investigator.
Time Frame: Baseline up to 28 days after last dose of study drug (up to 22 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Duavive
Number analyzed (Participants) | 639
Participants
  Treatment Related AEs | 58
  Treatment Related SAEs | 0

3. Primary Outcome: Number of Participants Classified According to Measures Taken for Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Following measures were taken for AEs in relation to Duavive tablet: no change in treatment, permanently discontinued treatment and temporarily discontinued treatment.
Time Frame: Baseline up to 28 days after last dose of study drug (up to 22 months)
Population: Safety analysis set included those participants who had been administered with Duavive tablet at least once and had completed follow up. Here, "Overall Number of Participants Analyzed" signifies number of participants with adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Duavive
Number analyzed (Participants) | 73
Participants
  No change in treatment | 19
  Permanently discontinued treatment | 53
  Temporarily discontinued treatment | 1

4. Primary Outcome: Number of Participants With Change From Baseline in Moderate to Severe Vasomotor Symptoms Associated With Menopause at Month 3
Description: Change from baseline in moderate to severe vasomotor symptoms associated with menopause was judged by investigator based on recorded symptoms and classified as "Effectiveness" when symptoms improved and as "Ineffectiveness" when there was no change in symptoms or symptoms aggravated.
Time Frame: Baseline, Month 3
Population: Efficacy analysis set (EAS) of treatment for moderate to severe vasomotor symptoms associated with menopause included those participants who were administered with Duavive tablet at least once and completed follow up and were evaluated for treatment of moderate to severe vasomotor symptoms associated with menopause. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure at Month 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Duavive
Number analyzed (Participants) | 387
Participants
  Effectiveness | 319
  Ineffectiveness | 68

5. Primary Outcome: Number of Participants With Change From Baseline in Moderate to Severe Vasomotor Symptoms Associated With Menopause at Month 6
Description: as for outcome 4
Time Frame: Baseline, Month 6
Population: EAS of treatment for moderate to severe vasomotor symptoms associated with menopause included those participants who were administered with Duavive tablet at least once and completed follow up and were evaluated for treatment of moderate to severe vasomotor symptoms associated with menopause. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure at Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Duavive
Number analyzed (Participants) | 141
Participants
  Effectiveness | 118
  Ineffectiveness | 23

6. Primary Outcome: Percentage of Participants With Improvement From Baseline in Moderate to Severe Vasomotor Symptoms Associated With Menopause at Last Visit
Description: Improvement from baseline in moderate to severe vasomotor symptoms associated with menopause was judged by investigator based on recorded symptoms and classified as "Effectiveness" when symptoms improved.
Time Frame: Baseline, Last visit (last visit was anytime up to a maximum of Month 21)
Population: EAS of treatment for moderate to severe vasomotor symptoms associated with menopause included those participants who were administered with Duavive tablet at least once and completed follow up and were evaluated for treatment of moderate to severe vasomotor symptoms associated with menopause.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Duavive
Number analyzed (Participants) | 390
percentage of participants | 82.31 [78.15 to 85.97]

7. Primary Outcome: Number of Participants With Prevention of Post-menopausal Osteoporosis at Month 3
Description: Investigator evaluated preventive effect of Duavive treatment based on comparing results of following at baseline and specified visit: X-ray examination, bone density test record, other blood test record related to resorption of bone and osteogenesis. In this outcome measure, data of only those participants in which Duavive treatment was effective in prevention of post-menopausal osteoporosis is reported.
Time Frame: Month 3
Population: EAS of prevention of postmenopausal osteoporosis included those participants who were administered with Duavive tablet at least once and completed follow up and were evaluated for prevention of post-menopausal osteoporosis.
Measure: Count of Participants; unit: Participants
Arm/Group | Duavive
Number analyzed (Participants) | 22
Participants | 17

8. Primary Outcome: Number of Participants With Prevention of Post-menopausal Osteoporosis at Month 6
Description: as for outcome 7
Time Frame: Month 6
Population: EAS of prevention of postmenopausal osteoporosis included those participants who were administered with Duavive tablet at least once and completed follow up and were evaluated for prevention of post-menopausal osteoporosis. Here, "Overall number of participants analyzed" = participants who were administered with Duavive tablet for prevention of postmenopausal osteoporosis at Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Duavive
Number analyzed (Participants) | 1
Participants | 1

9. Primary Outcome: Percentage of Participants With Prevention of Post-menopausal Osteoporosis at Last Visit
Description: as for outcome 7
Time Frame: Last visit (last visit was anytime up to a maximum of Month 21)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Duavive
Number analyzed (Participants) | 22
percentage of participants | 77.27 [54.63 to 92.18]

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (up to 22 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety analysis set.
Arm/Group | Duavive
All-Cause Mortality (participants affected / at risk) | 0/639
Serious Adverse Events (participants affected / at risk) | 2/639
Other Adverse Events (participants affected / at risk) | 71/639
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duavive (N=639)
Meniere's disease (Ear and labyrinth disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duavive (N=639)
Palpitations (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastric disorder (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Drug ineffective (General disorders) | 12
Face oedema (General disorders) | 3
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Genital herpes (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Weight increased (Investigations) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Flushing (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT02792504/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT02792504/SAP_001.pdf